CLINICAL TRIAL: NCT03337412
Title: Therapeutic Care and Education in Endocrinology-Diabetes-Nutrition: Evaluation of the Interest of the APA Educator (Adapted Physical Activity Educator) for the Establishment of Physical Activities in the Management and Prevention of Overweight and Obesity
Brief Title: Adapted Physical Activity Study
Acronym: APA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC16_0198
Record Dates: First submitted 2017-10-26; First posted 2017-11-09 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Obesity
Keywords: Therapeutic Education; physical activity; overweight; obesity
MeSH Terms: conditions — Obesity; Motor Activity; Overweight

STUDY DESIGN:
Intervention Model Description: uncontrolled, non-randomized, open-plan, multi-centre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): initial assessment of physical capacities, determination of personalized objectives on the occasion of 1 to 2 workshops during the hospital checkup. Telephone Contact by the APA educator at 6 months. One-year medical visit.
  Interventions: Other: Adapted physical activity
- Employees (Experimental): initial assessment of physical capacities, participation in 10 to 20 physical activity workshops over 6 months on working time, then employees oriented towards autonomous activities over the following 6 months.
  Evaluation by computer-filled questionnaires.
  Interventions: Other: Adapted physical activity

INTERVENTIONS:
Other: Adapted physical activity — Patients will be asked to complete questionnaires about their physical activity, diet and quality of life prior to hospital care.For an evaluation of the chronological evolution of their physical activity, they will be invited to complete the Physical Activity Questionnaire GPAQ 2.0 every 2 months, for the duration of the Research.At 6 months during a telephone contact and at 12 months, during a consultation, the food and quality of life questionnaires will also have to be informed. The evolution of weight, body mass index and metabolic biological factors will also be collected.
  Employees will benefit from a life-health awareness program, accompanied by an APA educator, they are offered the opportunity to participate in physical activity workshops on a regular basis (12 workshops minimum over 6 months), adapted to their abilities and personalized.They will be invited to fill, from their home or on the website Fleury Michon, the same type of questionnaire

SUMMARY:
An uncontrolled, non-randomized, open-plan, multi-centre study of treatment and therapeutic education in endocrinology-diabetes-Nutrition that seeks to assess the interest of an adapted physical activity educator for the implementation In place of physical activities in the management and prevention of overweight and obesity. The proposed study seeks to promote the physical activity (PA) to patients and employees, including the encouragement of physical activity in a guided and personalized way, through workshops on working time, and follow-up of the evolution of the PA through a Adapted questionnaire.

DETAILED DESCRIPTION:
The evaluation will be proposed

* in the Department of Endocrinology, Metabolic diseases and Nutrition of the Nantes University Hospital to all patients participating in "overweight education groups" in complete hospitalization or in day hospital
* to the employees of the group Fleury-Michon volunteers.
* During a recruitment period of 6 months required for the recruitment of 100 patients and 80 employees;
* For a total duration of the research for each 1 year participant. Patients and employees will be systematically informed of the project and their consent will be collected by oral and plotted in the medical file and in the employee file, kept by the adapted physical activity educator.

For the hospital phase, patients will be asked to complete questionnaires regarding their physical activity, diet and quality of life prior to hospital care. For an evaluation of the chronological evolution of their physical activity, they will be invited to complete the global Physical Activity Questionnaire (GPAQ 2.0), every 2 months, from their home, via the Internet from a secure link (ECRF clinsight) for the duration of the Research is one year. At 6 months during a telephone contact and at 12 months, during a consultation, the food and quality of life questionnaires will also have to be informed. The evolution of weight, body mass index (BMI) and metabolic biological factors (fasting blood glucose and lipid balance) will also be collected.

For the enterprise phase, employees will benefit from a life-health awareness program, accompanied by an APA educator, they are offered the opportunity to participate in physical activity workshops on a regular basis (12 workshops minimum over 6 months), adapted to their abilities and personalized. They will be invited to fill, from their home or on the website Fleury Michon, via the Internet from a secure link (ECRF clinsight) the same type of questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients hospitalized for weight problem in the service of endocrinology, metabolic diseases and Nutrition of the Nantes University Hospital's and employees of the company Fleury-Michon not contraindicated to the practice of a sports activity by the dealing doctor
* benefiting from the intervention of an APA educator
* able to complete the questionnaires of physical activity, eating habits, quality of life and satisfaction
* having given their oral consent

Exclusion Criteria:

* Major subjects protected, under guardianship or curators;
* Pregnant women on a declarative test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Chronological evolution of the physical activity score of patients benefiting from the education program with intervention of the adapted physical activity educator | every 2 months over 12 months
  Physical activity will be evaluated both qualitatively (low, moderate and intense) and quantitatively (expressed as metabolic Equivalent of Task: MET-min/week) through the World Health Organization GPAQ 2.0 questionnaire, based on physical activities at work, In moving and hobbies.

SECONDARY OUTCOMES:
Changes in eating habits | at 6 months and 1 year
  simple questionnaire on food groups consumed
Evolution of BMI | at 6 months and 1 year
Evolution of the basic energy expenditure | at 12 months
  evaluated by calorimetry or impedance
Evolution of metabolic parameters (fasting blood glucose and lipid balance) | at 12 months
  fasting blood glucose and lipid balance are measured systematically for patients with hospital care, and are optional according to the biological balances already performed for the employees
Evolution of the quality of life | at 6 months and 1 year
  Short Form 36 (SF36) Questionnaire
Evolution of patients satisfaction | at 6 months and 1 year
  specific questionaire
musculoskeletal disorders | at 6 months and 1 year
  For employees will also be evaluated certain specific indicators of occupational diseases such as musculoskeletal disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Marie GUILLOUCHE, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No